CLINICAL TRIAL: NCT04030195
Title: A Phase 1/2a, Open-label, Dose-escalation, Dose-expansion, Parallel Assignment Study to Evaluate the Safety and Clinical Activity of PBCAR20A in Subjects With Relapsed/Refractory (r/r) Non-Hodgkin Lymphoma (NHL) or r/r Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Dose-escalation Study of Safety of PBCAR20A in Subjects With r/r NHL or r/r CLL/SLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precision BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBCAR20A-01
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Non-Hodgkin's Lymphoma, Relapsed; Chronic Lymphoid Leukemia in Relapse; Non-Hodgkin's Lymphoma Refractory; Chronic Lymphocytic Leukemia; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic; B-cell Chronic Lymphocytic Leukemia; B-cell Non Hodgkin Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Phase 1: Participants with r/r CD20+ B-cell NHL or r/r CLL/SLL will be enrolled to 3 escalating dose groups and treated sequentially, with the possibility of a single de-escalation. Within each dose group, at least 3 and at most 6 study participants will be treated with a single dose of PBCAR20A using a standard 3 + 3 design. The starting dose of PBCAR20A will be 1 × 10^6 chimeric antigen receptor (CAR) T cells/kg body weight. Subsequent dose groups will be treated with escalating doses to a maximum dose of 480 × 10^6 CAR T cells (flat dose). In the absence of dose-limiting toxicities (DLTs) (as described in Section 3.8 of the protocol), the dose will be increased using a fixed-dose scheme.
  Phase 2: Study PBCAR20A-01 did not proceed into Phase 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 of PBCAR20A CAR T cells (Experimental): 1 x 10^6 chimeric antigen receptor (CAR) T cells per kg body weight.
  In this study, PBCAR20A, allogeneic anti-cluster of differentiation (CD20) CAR T Cells, is used to treat patients with relapsed or refractory (r/r) CD20+ Non-Hodgkin Lymphoma (NHL) or r/r Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL).
  Route of Administration: Intravenous infusion (IV)
  Lymphodepletion Conditioning: Lymphodepletion will be conducted several days prior to PBCAR20A infusion. A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Genetic: PBCAR20A; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 2 of PBCAR20A CAR T cells (Experimental): 240 x 10^6 CAR T cells (flat dose)
  Interventions: Genetic: PBCAR20A; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 3 of PBCAR20A CAR T cells (Experimental): 480 x 10^6 CAR T cells (flat dose)
  Interventions: Genetic: PBCAR20A; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: PBCAR20A — Single dose of Allogeneic Anti-CD20 CAR T cells will be infused, and a classic "3+3" dose escalation will be applied.
  Other Names: Allogeneic Anti-CD20 CAR T cells
Drug: Fludarabine — Fludarabine is used for lymphodepletion (30 mg/m^2/day, Days -5 to -3).
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion (500 mg/m^2/day, Days -5 to -3).

SUMMARY:
This is a Phase 1/2a, nonrandomized, open-label, parallel assignment, single-dose, dose-escalation, and dose-expansion study to evaluate the safety and clinical activity of PBCAR20A in adult subjects with r/r B-cell NHL or r/r CLL/SLL.

DETAILED DESCRIPTION:
This is a multicenter, nonrandomized, open-label, parallel assignment, single-dose, dose-escalation, and dose-expansion study to evaluate safety, tolerability, clinical activity, and find an appropriate dose to optimize safety and efficacy of PBCAR20A in subjects with relapsed/refractory (r/r) CD20+ Non-Hodgkin Lymphoma (NHL) or r/r Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL). Before initiating PBCAR20A, therapy, subjects will be administered lymphodepletion chemotherapy composed of fludarabine and cyclophosphamide. At Day 0 of the Treatment Period, subjects will receive a single intravenous (IV) infusion of PBCAR20A. All subjects are monitored during the treatment period through Day 28. All subjects who receive a dose of PBCAR20A will be followed in a separate long-term follow-up (LTFU) study for 15 years after exiting this study.

ELIGIBILITY:
Key Inclusion Criteria

Criteria for NHL:

* r/r CD20+ B-cell NHL that is histologically confirmed by archived tumor biopsy tissue from the last relapse and corresponding pathology report.
* Measurable or detectable disease according to the Lugano classification.
* Primary refractory disease or r/r disease after a response to 2 prior regimens.

Criteria for CLL/SLL:

* Diagnosis of CD20+ CLL with indication for treatment based on the iwCLL guidelines and clinically measurable disease or SLL with measurable disease that is biopsy-proven SLL.
* Previously failed/tolerant to at least 2 prior lines of systemic targeted therapy of known benefit.

Criteria for both NHL and CLL/SLL:

* Study participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Study participant has adequate bone marrow, renal, hepatic, pulmonary, and cardiac function.

Key Exclusion Criteria:

Criteria for NHL:

* Requirement for urgent therapy due to mass effects such as bowel obstruction, spinal cord, or blood vessel compression.
* Active central nervous system (CNS) disease. A negative computed tomography (CT)/magnetic resonance imaging (MRI) is required at Screening if the study participant has a history of CNS lymphoma.

Criteria for NHL and CLL/SLL:

* Active CNS disease. A negative lumbar puncture is required at Screening if the study participant has a history of CNS disease.
* Previous malignancy, besides the malignancies of inclusion (B-cell NHL or CLL/SLL), that in the investigator's opinion, has a high risk of relapse in the next 2 years.
* Active uncontrolled fungal, bacterial, viral, protozoal, or other infection.
* Any form of primary immunodeficiency.
* History of human immunodeficiency virus (HIV) infection.
* Active hepatitis B or C.
* Uncontrolled cardiovascular disease.
* Hypertension crisis or hypertensive encephalopathy within 3 months prior to Screening.
* Presence of a CNS disorder that renders ineligible for treatment.
* History of a genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman Diamond syndrome, or any other known bone marrow failure syndrome.
* Received ASCT within 45 days of Screening if the study participant has met the rest of the count requirements.
* Must not have received systemic corticosteroid therapy for at least 7 days prior to initiating lymphodepletion chemotherapy.
* Received a live vaccine within 4 weeks before Screening.
* Radiotherapy within 4 weeks determined on a case-by-case basis.
* Presence of a pleural/peritoneal/pericardial catheter.
* Current use of any anticoagulant or antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan List, MD, Study Chair — Precision BioSciences, Inc.
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Stanford University, Stanford, California
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants were screened for this study, of whom 2 screen failed.
Groups:
- Dose Level 1 of PBCAR20A CAR T Cells: 1 x 10^6 CAR T cells per kg body weight.
  In this study, PBCAR20A, allogeneic anti-CD20 CAR T Cells, is used to treat patients with relapsed or refractory (r/r) Non-Hodgkin Lymphoma (NHL) or r/r Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL).
  Route of Administration: Intravenous infusion.
  Lymphodepletion Conditioning: Lymphodepletion will be conducted several days prior to PBCAR20A infusion. A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  PBCAR20A: Single dose of Allogeneic Anti-CD20 CAR T cells will be infused, and a classic "3+3" dose escalation will be applied.
  Fludarabine: Fludarabine is used for lymphodepletion (30 mg/m^2/day, Days -5 to -3).
  Cyclophosphamide: Cyclophosphamide is used for lymphodepletion (500 mg/m^2/day, Days -5 to -3).
Period: Overall Study
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells
Started (One participant who was retreated was dosed with Dose Level 3 at both initial and retreatment dosing. For the purposes of calculating and reporting participant flow and efficacy outcomes, the participant who was dosed twice was counted as 2 individual participants.) | 8 | 3 | 7
Participants in Demographic Population | 8 | 3 | 6
Participants in Safety Population | 8 | 3 | 6
Participants Re-treated | 0 | 0 | 1
Participants in Efficacy Population | 8 | 3 | 7
Completed | 6 | 3 | 7
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 of PBCAR20A CAR T Cells: 1 x 10^6 CAR T cells per kg body weight
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells | Total
Number analyzed (Participants) | 8 | 3 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.25 (17.07) | 47.00 (19.08) | 58.17 (13.70) | 56.24 (15.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 6 | 3 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 7 | 1 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 2 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD) is the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT) using a 3+3 strategy.
Time Frame: Day 1 to Day 28
Population: All participants. The participant who was dosed twice at Dose Level 3 (DL3) was counted as 2 individual participants.
Measure: Number; unit: 10^6 CAR T cells
Groups:
- PBCAR20A CAR T Cells: All participants who received PBCAR20A CAR T Cells at any dose level
Arm/Group | PBCAR20A CAR T Cells
Number analyzed (Participants) | 18
10^6 CAR T cells | NA — MTD was not reached in this study because MTD requires at least 2 dose limiting toxicities (DLTs) in any given dose level and only 1 DLT was noted.

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: Dose-limiting toxicities (DLT) are certain Grade 3 and Grade 4 toxic reactions as defined by the protocol and CTCAE v5.0.
Time Frame: 1 year
Population: All participants. The participant who was dosed twice at DL3 was counted as 2 individual participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells
Number analyzed (Participants) | 8 | 3 | 7
Participants | 1 | 0 | 0

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is a measure of clinical activity as response in NHL by the revised Lugano Classification (Cheson et al, 2016) or a response in CLL/SLL by the International Workshop on Chronic Lymphocytic Leukemia 2018 guidelines.
Time Frame: 1 year
Population: All participants. The participant who was dosed twice at DL3 was counted as 2 individual participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells
Number analyzed (Participants) | 8 | 3 | 7
Participants
  Responders | 2 | 1 | 3
  Complete Response | 1 | 0 | 0
  Partial Response | 1 | 1 | 3
  Non-responders | 6 | 2 | 4

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration (days) from Day 0 to disease progression or death.
Time Frame: 1 year
Population: All participants. The participant who was dosed twice at DL3 was counted as 2 individual participants.
Measure: Median (Full Range); unit: Days
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells
Number analyzed (Participants) | 8 | 3 | 7
Days | 29.5 [15.0 to 365.0] | 29.0 [29.0 to 94.0] | 29.0 [12.0 to 66.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1 of PBCAR20A CAR T Cells | Dose Level 2 of PBCAR20A CAR T Cells | Dose Level 3 of PBCAR20A CAR T Cells
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 of PBCAR20A CAR T Cells (N=8) | Dose Level 2 of PBCAR20A CAR T Cells (N=3) | Dose Level 3 of PBCAR20A CAR T Cells (N=6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
CAR T cell-related encephalopathy syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 of PBCAR20A CAR T Cells (N=8) | Dose Level 2 of PBCAR20A CAR T Cells (N=3) | Dose Level 3 of PBCAR20A CAR T Cells (N=6)
Anaemia (Blood and lymphatic system disorders) | 6 (13) | 1 (1) | 3 (8)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (6) | 2 (4) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 4 (7)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 2 (4) | 3 (6)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (1) | 3 (3)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (11) | 2 (3) | 4 (10)
Platelet count decreased (Investigations) | 3 (4) | 0 (0) | 3 (7)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (6) | 1 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 2 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
CAR T-cell-related encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 2 (4) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT04030195/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04030195/SAP_001.pdf